CLINICAL TRIAL: NCT05804942
Title: Metabolic Response to Variations in Dietary Glycemic Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Chief scientist, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SIAT-IRB-221115-H0618
Record Dates: First submitted 2023-02-17; First posted 2023-04-07 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Hunger; Food Preferences
Keywords: carbohydrate insulin model; circulating factors
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High glycemic index (Experimental): The participants will be fed a fixed calorie meal, which is high glycemic index with constant fat and protein.
  Interventions: Behavioral: High glycemic index
- Medium glycemic index (Experimental): The participants will be fed a fixed calorie meal, which is medium glycemic index with constant fat and protein.
  Interventions: Behavioral: Medium glycemic index
- Low glycemic index (Experimental): The participants will be fed a fixed calorie meal, which is low glycemic index with constant fat and protein.
  Interventions: Behavioral: Low glycemic index

INTERVENTIONS:
Behavioral: High glycemic index — Composition (by proportion of calories) of meal: 60% carbohydrate (glycemic index:>70), 20% fat and 20% protein.
  Arms: High glycemic index
Behavioral: Medium glycemic index — Composition (by proportion of calories) of meal: 60% carbohydrate (glycemic index:55-70), 20% fat and 20% protein.
  Arms: Medium glycemic index
Behavioral: Low glycemic index — Composition (by proportion of calories) of meal: 60% carbohydrate (glycemic index:<55), 20% fat and 20% protein.
  Arms: Low glycemic index

SUMMARY:
The goal of this study is to compare metabolic response to variations in dietary glycemic index in healthy participants. The main questions it aims to answer are:

• What are the metabolic hunger and food intake responses to different levels of glycemic index on the background of otherwise constant macronutrient composition? Participants will come to the lab after an overnight fast and body composition will be tested by bio-impedance analysis and magnetic resonance imaging. They will then be randomized to eat one of three standardized breakfasts varying in the glycemic index. Circulating glucose levels will be monitored using a continuous glucose monitor and blood samples will be collected to measure metabolic and hormone factors in the serum. Participants will also rate their hunger at 0, 30, 60, 120, 180, 240 and 300 minutes. After 5 hours they will eat a free choice meal from a standardized selection buffet (test meal).

DETAILED DESCRIPTION:
The primary variable in this study is the food energy intake at the test meal consumed 5 hours after the dietary intervention meal on day1 of the experiment, compared to the intake of the same test meal consumed on day 0. The investigators performed a power analysis using this outcome measure to inform the sample size if the data were analysed using one-way ANOVA. The number of levels in the study is 3, the investigators set the effect size as a difference between means of the groups of 265 kJ. From a pilot study of repeated measurements across individuals the investigators observed the standard deviation of the difference between repeated intakes was 372 kJ. The investigators set the power value of the study at 80 %. This analysis suggested a sample of 39 individuals per group. To account for individuals potentially not completing the study, the investigators aimed to recruit 135 participants in total.

The experiment includes the pre-test, the dietary intervention and postprandial monitoring.

Pre-test. The participants will be fed a test meal (free choice from buffet) at noon the day before the experiment (day 0). The food preference and total energy intake will be assessed. On the experimental day (day 1), the participants will be asked to attend the laboratory in the morning after an overnight fast (10 hours fasting). The body composition will be measured using a bio-impedance and magnetic resonance imaging, Then the participants will be guided to wear a continuous glucose monitoring system (CGMS) and the CGMS is under initialization for 2 hours. Also, a peripheral venous catheter (PVC) will be placed in the back of the hand, upper arm or elbow socket and 6 ml of fasting peripheral blood will be drawn (0 min).

Dietary intervention. 60 male and 60 female participants will be randomly divided into three groups: low, moderate and high glycemic index groups. Each group consists of 20 males and females. They will be feed by standardized meal with constant fat, protein and carbohydrate % but differing in the source of the carbohydrates.

Postprandial test. The test includes the testing of physiological indices during and after the intervention meal. In addition to continuously recording the changes in blood glucose by CGMS, the hunger rate will be accessed at 30 minutes intervals and peripheral blood will be collected by PVC (6 ml each time) at 30, 60, 120, 180, 240 and 300 min after the meal. When the participants have finished the tests during 300 min, a test meal will be provided identical to that provided on day 0. The effect of the standard meal on the total energy intake and macronutrient (carbohydrate, protein, fat) supply will be accessed in absolute amounts and the change between day 0 and day 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (both men and women)
* 18-40 years old
* 18.5 ≤ BMI (body mass index)<24 kg/m2

Exclusion Criteria:

* Those who have undergone surgery in the past 6 months.
* People are requiring long-term medication.
* People have metabolic diseases, like diabetes, hypoglycemia, gout, osteoporosis, et al.
* Those who have recently lost weight for various medical reasons (e.g. cancer, etc.).
* People are losing weight by tablets.
* People are suffering from infectious diseases (e.g. HIV, etc.)
* People have blood phobia, pathological hypo or hyper tension.
* People with impaired glucose tolerance.
* Pregnant and lactation women.
* Those who are afflicted with claustrophobia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in energy intake of test meal between day 0 and day 1 | Change in intake between day 0 and day 1
  The food intake will be assessed objectively by use of a feeding table. The test meal will be provided as lunch, and food types available on the table include staples, vegetables, mushrooms, meat, soy products, desserts, beverages and water. All types of food are unlimited. Food consumption will be recorded continuously by balances concealed under each food dish. The food energy density for each food will be measured by bomb calorimetry in kJ/g, and energy intake will be calculated as the product of the grams of each food eaten multiplied by the respective energy density and then summed, as kJ.
  This test meal intake is measured on day 0 and then a repeat test meal measure is made under identical conditions on day 1. On day 1 an intervention meal is also consumed five hours before the test meal is consumed. On day 0 no such meal is consumed. The outcome measure is the change in food intake (kJ) between day 0 and day 1 reflecting the impact of the intervention meal.

SECONDARY OUTCOMES:
circulating hormones | fasting, postprandial 30, 60, 120, 180, 240 and 300 minutes.
  Nurses will collect the blood samples on day 1. Levels of circulating hormones (insulin, leptin, glycogen,etc) in the serum will be measured by ELISA(Bio Tek, Synergy4) in mmol/L.
postprandial glucose | fasting glucose and postprandial glucose for 5 hours
  Standardized meal with different levels of glycemic index( low level: ≤ 55, moderate level: 55 < GI ≤ 70, high level: > 70) will be provided as breakfast on day 1. Independent of the GI, the energy supply ratio of macronutrients carbohydrate, protein and fat will be fixed at 60 %, 20 % and 20 % respectively. Glucose concentration after the standardized meal will be recorded by the continuous glucose monitoring system(Medtronic) in mmol/L during 5 hours.
self reported hunger | fasting, postprandial 30, 60, 120, 180, 240 and 300 minutes.
  Self reported hunger will be tested by rating scale question.
levels of circulating metabolic fuels | fasting, postprandial 30, 60, 120, 180, 240 and 300 minutes.
  Nurses will collect the blood samples on day 1. Circulating lactate, free-fatty acids, triglycerides etc in mmol/L will be measured by ELISA(Bio Tek, Synergy4).

OTHER OUTCOMES:
fat mass tested by bioelectrical impedance analysis | pre measurement
  Fat mass will be tested by bioelectrical impedance analysis(Tanita, MC-980) in kg.
fat mass tested by magnetic resonance imaging | pre measurement
  Fat mass will be tested by magnetic resonance imaging(Shanghai united imaging, uMR790) in %.
fat free mass tested by bioelectrical impedance analysis | pre measurement
  Fat free mass will be tested by bioelectrical impedance analysis(Tanita, MC-980) in kg.
fat free mass tested by magnetic resonance imaging | pre measurement
  Fat free mass will be tested by magnetic resonance imaging(Shanghai united imaging, uMR790) in %.
sex difference in energy intake | pre measurement
  The impact of sex on energy intake will be explored by correlation analysis.
sex difference in circulating hormones | pre measurement
  The impact of sex on circulating hormones will be explored by correlation analysis.
sex difference in postprandial glucose | pre measurement
  The impact of sex on postprandial glucose will be explored by correlation analysis.
sex difference in self reported hunger | pre measurement
  The impact of sex on self reported hunger will be explored by correlation analysis.
sex difference in circulating metabolic fuels | pre measurement
  The impact of sex on circulating metabolic fuels will be explored by correlation analysis.
sex difference in fat mass | pre measurement
  The impact of sex on fat mass will be explored by correlation analysis.
sex difference in fat free mass | pre measurement
  The impact of sex on fat free mass will be explored by correlation analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Institutes of Advanced Technology, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No